CLINICAL TRIAL: NCT05501964
Title: Predictors and Outcomes of Time to Hemostasis Post Trans-femoral Cardiac Catheterization: a Multicenter Cohort Study
Brief Title: Predictors and Outcomes of Time to Hemostasis After Cardiac Catheterization
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Maha Gamal Ramadan Asal, Principle investigator, Alexandria University
Other Study IDs: 1552022
Record Dates: First submitted 2022-08-06; First posted 2022-08-16 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to:

1. Assess the incidence of hemostasis failure after manual compression of trans-femoral arterial sheath post percutaneous coronary intervention.
2. Assess the predictors of time to hemostasis achieved by manual compression for trans-femoral arterial sheath post percutaneous coronary intervention.
3. Assess the association between time to hemostasis and the incidence of vascular access complications after manual compression for trans-femoral arterial sheath removal post percutaneous coronary intervention.
4. Assess the association between failed hemostasis and the incidence of vascular access complications after manual compression for trans-femoral arterial sheath removal post percutaneous coronary intervention.

DETAILED DESCRIPTION:
Nurses and medical professionals have a vital role in detecting, preventing, and managing complications at the earliest possible stage. They should assess patients for high risk of complications, and plan management strategies to decrease those complications. In many acute and critical care settings, removing femoral sheaths and handling related complications after percutaneous coronary intervention. are primarily the responsibilities of nurses. Therefore, after catheterization procedures, assessing the predictors of required time to achieve optimal hemostasis at the time of trans-femoral arterial sheath removal is essential as one of the final modifiable measures to prevent access site complications. This study will be done in 6 Cardiac catheterization units representing governmental and private hospitals. A sample size of 266 patients will be recruited for the study. data will be analyzed by univariate and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who planned for elective or primary percutaneous coronary intervention with femoral access, and
* Agreed to participate in the study

Exclusion Criteria:

* Patients who had trans-femoral catheterization procedure within a 1-month duration
* patients with a known history of coagulation disorders,
* patients with sheath removed at the laboratory, and
* Patients who experience post - catheterization life-threatening events rather than vascular access complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample size of 266 percutaneous coronary intervention patients is needed to detect the rate of complications after manual compression. Assuming the rate of complications according to a previous study was 4%, with an assumed population proportion of 8% using a two-sided, binomial hypothesis test with a target significance level of 0.05.
  Also, the sample size is sufficient to assess the meantime to homeostasis (26±15) min, with a precision of 4 min, according to a previous study, at a significance level of .05, using the One-sample t-test. The sample size was calculated using NCSS 2004 and PASS 2000 software.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2024-05-05 (Actual)

PRIMARY OUTCOMES:
Time to hemostasis | 12 hours after percutaneous coronary intervention
  The time frame (minutes) required for manual compression from the removal of sheath to achieve hemostasis
Pre-procedure predictor factors associated with change of the mean time to hemostasis | before percutaneous coronary intervention
  Patient and procedure-related factors will be assessed by patient demographics and clinical data questionnaire. This questionnaire will gather data regarding patient demographics, comorbidities, risk factors, blood chemistry medications taken, and angiographic factors that can predict the mean time to safe hemostasis.
Intra-procedure- predictor factors associated with a change in the mean time to hemostasis | during percutaneous coronary intervention
  Intra-procedure factors as measured by the percutaneous coronary intervention factors assessment checklist. This checklist will gather data regarding, puncture site, the number of punctures, guiding Catheter size, medications taken, procedure duration, amount of dye used, fluoroscopy time and the procedure done, and years of operator experience. These factors will be analyzed using multiple regression to identify intra-procedure predictor factors associated with a change in the mean hemostasis time.
Trans-Femoral Arterial Sheath Removal Predictor factors associated with a change in the mean time to hemostasis | 12 hours after percutaneous coronary intervention "during arterial sheath removal"
  Trans-Femoral Arterial Sheath Removal Variables checklist. This checklist gathers data regarding sheath removal time after the procedure, heart rate, and blood pressure before and after sheath removal, failed closure, ambulation time after sheath removal qualification, and years of experience of the health care provider who removes the sheath. These factors will be analyzed using multiple regression to identify trans-femoral arterial sheath removal factors associated with a change in the mean hemostasis time.
Rate of the vascular Access Complications occurrence | 12 hours after percutaneous coronary intervention "during arterial sheath removal"
  Complication rate as assessed by the number of events for oozing, ecchymosis, hematoma, bleeding, pseudoaneurysm, arteriovenous fistula, and femoral occlusion as assessed by the assigned nurse and treating physician
Rate of the vascular Access Complications occurrence | 6 hours after sheath removal
  Complication rate as assessed by the number of events for oozing, ecchymosis, hematoma, bleeding, pseudoaneurysm, arteriovenous fistula, and femoral occlusion as assessed by the assigned nurse and treating physician
Rate of the vascular Access Complications occurrence | 12 hours after sheath removal
  Complication rate as assessed by the number of events for oozing, ecchymosis, hematoma, bleeding, pseudoaneurysm, arteriovenous fistula, and femoral occlusion as assessed by the assigned nurse and treating physician
Rate of the vascular Access Complications occurrence | immediately before patient discharge from the hospital
  The complication rate will be assessed by the number of events for oozing, ecchymosis, hematoma, bleeding, pseudoaneurysm, arteriovenous fistula, and femoral occlusion as assessed by the assigned nurse and treating physician.

SECONDARY OUTCOMES:
Groin pain | Immediately after femoral sheath removal
  Severity of the pain experienced by the patient as assessed by the pain Visual Analog Scale. the scale score range from 0-10. score of 0 indicate "no pain", 1-3 " mild pain", 4-6 "moderate pain", and 7-10 " severe pain"

CONTACTS AND LOCATIONS:
Overall Officials: Maha G Asal, Phd, Principal Investigator — Alexandria University; Eshrak S Hashem, Phd, Principal Investigator — Alexandria University; Wafaa H Awad, Phd, Principal Investigator — Alexandria University
Locations (5):
- Egypt (5):
  - Andalusia Private Hospital, Alexandria
  - German Heart Center, Alexandria
  - Mabaret Aalsafra hospital, Alexandria
  - Shark El-Madina Hospital, Alexandria
  - Smouha University hospital, Alexandria

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make individual participant data available.